CLINICAL TRIAL: NCT06096649
Title: Prospective Randomized Vehicle-Controlled Double-Blind Assessment of the Effects of Zinc Di-(Dibutyryl Lisinate) on Skin Biophysical Properties and the Skin Microbiome in Photoaged Skin
Brief Title: The Effects of Zinc Di-(Dibutyryl Lisinate) on Skin Health and the Skin Microbiome in Photoaged Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Sytheon Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: i23-08-ZBL-SYTH
Record Dates: First submitted 2023-10-12; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Photoaging
Keywords: skin microbiome; skin biophysical properties; photoaging; zinc di-(dibutyryl lisinate)

STUDY DESIGN:
Intervention Model Description: Zinc Di-(dibutyryl lisinate) vs Vehicle
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Vehicle + Zinc Di-(dibutyryl lisinate) (Experimental): Topical cream containing Zinc Di-(dibutyryl listinate)
  Interventions: Other: Topical Vehicle + Zinc Di-(dibutyryl lisinate)
- Topical Vehicle (Placebo Comparator): Topical cream
  Interventions: Other: Topical Vehicle

INTERVENTIONS:
Other: Topical Vehicle + Zinc Di-(dibutyryl lisinate) — Instructions: Apply to the entire face twice daily - morning and evening
  Arms: Topical Vehicle + Zinc Di-(dibutyryl lisinate)
Other: Topical Vehicle — Instructions: Apply to the entire face twice daily - morning and evening
  Arms: Topical Vehicle

SUMMARY:
This study is a double-blind randomized vehicle-controlled study assessing how Zinc Di-(dibutyryl lisinate) (Z-DBL) influences skin biophysical measures such as skin hydration, transepidermal water loss, and elasticity, as well as its effects on the skin microbiome of photoaged skin.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 40 years of age until 60 years of age
* Participants must have facial fine lines and wrinkles
* Subjects must minimize sun exposure
* Subjects must avoid professional or facial spa procedures during the study

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners.
* Adults unable to consent.
* Those who are unwilling to discontinue topical hydroquinone, retinoids, bakuchiol, vitamin C, or acetyl zingerone containing products for two weeks to meet the washout criteria prior to enrolling.
* Those who are unwilling to discontinue topical antibiotics and benzoyl peroxide for two weeks to meet the washout criteria prior to enrolling.
* Those who have been on an oral antibiotic within 1 month prior to enrolling.
* Subjects with any of the following facial cosmetic treatments in the past 3 months or those who are unwilling to withhold the following facial cosmetic treatments during the study including botulinum toxin, injectable fillers, microdermabrasion, intense pulsed light (IPL), peels, laser treatments, acid treatments, facial plastic surgery, or any other medical treatment administered by a physician or skin care professional which is designed to improve the appearance of facial skin.
* Those who are unwilling to discontinue all facial topical products except the product provided in the study.
* Individuals who have changed any of their hormonal based contraception within 3. months prior to joining the study.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in image analysis based pigment intensity | 8 weeks
  Facial photographs will be analyzed for pigment intensity for the face after the photographs are obtained and analyzed utilizing the BTBP 3D Clarity Pro Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA, USA). The pigment intensity will be measured as a relative change from baseline and is a dimensionless and normalized measure.
Skin Hydration | 8 weeks
  The skin capacitance will be measured with a handheld non-invasive device (Skin MoistureMeterSC, Delfin Technologies Ltd.). The measurement is in arbitrary units per manufacturer.

SECONDARY OUTCOMES:
Change in image analysis based wrinkle severity | 8 weeks
  Facial photographs will be obtained and analyzed utilizing the BTBP 3D Clarity Pro Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA, USA). The measurement will analyze wrinkle severity that is a measure of both the wrinkle depth and width and will be reported as a relative change from baseline.
Shifts in the skin microbiome diversity | 8 weeks
  Whole genome sequencing of the skin microbiome
Changes in skin barrier biomarkers like filaggrin | 8 weeks
  Measured using D-squame tape strips (CuDerm LLC.)
Product tolerability | 8 weeks
  Assessed with the use of a tolerability questionnaire to be completed by participants. Tolerability will be measured by rating symptoms such as burning, stinging, and scaling.
Change in skin elasticity | 8 weeks
  Skin elasticity measured with a handheld non-invasive device (Elastimeter, Delfin Technologies Ltd.)
Change in skin transepidermal water loss | 8 weeks
  Skin transepidermal water loss measured with a handheld non-invasive device (Vapometer, Delfin Technologies Ltd.)

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No